CLINICAL TRIAL: NCT02641262
Title: Henan ST-segment Elevation Myocardial Infarction (STEMI) Registry
Brief Title: Henan STEMI Registry
Status: Completed | Type: Observational
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Principal Investigator, Chuanyu Gao, Director, Henan Institute of Cardiovascular Epidemiology
Other Study IDs: HenanICE201501
Record Dates: First submitted 2015-12-15; First posted 2015-12-29 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: ST-segment Elevation Myocardial Infarction
Keywords: Myocardial Infarction; Angioplasty, Balloon, Coronary; Drug Therapy
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

SUMMARY:
ST-segment elevation myocardial infarction (STEMI) remains among the most acute and critical diseases, with primary percutaneous coronary intervention (pPCI) and thrombolysis as mainstay reperfusion treatments. Real-world implementation of current guidelines for STEMI management has been assessed in developed countries and large Chinese cities. However, until now, there has been no registry on patients with STEMI in Henan, the most populated (about 100 million) and predominantly rural (66%) province in central China.

This registry is aimed to assess management practices, time delays, outcomes and reasons for not receiving reperfusion therapy in consecutive STEMI patients in reperfusion-capable hospitals, i.e., tertiary and secondary, in Henan province.

DETAILED DESCRIPTION:
1. Henan institute of cardiovascular epidemiology is responsible for design, data quality control and statistical analysis.
2. Data are collected using a uniformed questionnaire by trained staff at each hospital.
3. Sample size estimation: Based on Henan retrospective observational cohort of STEMI patients, in-hospital mortality in secondary and tertiary hospitals were 5.6% and 6.0%, respectively. To achieve a precision of 20% with an α of 0.05 in each of the hospital, investigators need a sample of 5000, 2500 in each class hospital.
4. Statistical analysis plan: Investigators will report summary statistics for patient characteristics, delay time (symptom onset-to-first medical contact(FMC), FMC-to-reperfusion), patient referral (time and means of transportation), treatments received and primary outcomes. Investigators will also undertake the following prespecified subgroup analyses: hospital class, age, sex, killip class, time to first medical contact, infarct location, history of hypertension, diabetes or smoking and thrombolysis in myocardial infarction risk score.
5. Quality assurance plan

1)Diagnosis of STEMI is according to the third universal definition of myocardial infarction.

2)Before registry, a training program on study objectives, data collection, and STEMI management is given to the primary investigator and related staff at each participating center.

3)Henan institute of cardiovascular epidemiology will regularly monitored at least 10% of questionnaires for accuracy against medical records. If the questionnaires are not completed with 98% accuracy, all questionnaires are considered unqualified and this staff will be retrained.

4)Real-time automatic logic and range check on the completeness and validity of the data are integrated in the data entry system to control basic data quality. Henan ICE regularly provides data quality checks and sends queries for illogical, invalid or missing data elements to participating hospitals to review and revise. Participating centres who has the high error rate of data, and no change in 6 months shall be deemed abandoned automatically; participating centres who has the high quality of data will be issued a certificate to reward.

5)Investigator meeting will be annually held to conclude the progress, solve existing problems and strengthen program training.

ELIGIBILITY:
Inclusion Criteria:

* STEMI is defined in accordance with the universal definition of myocardial infarction, specifically as persistent ST-segment elevation (≥0.1 millivolt at J points) in 2 or more contiguous leads.

Exclusion Criteria:

* percutaneous coronary intervention (PCI)-related myocardial infarction or coronary artery bypass graft (CABG)-related myocardial infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STEMI patients within 30 days of symptom onset
Sampling Method: Probability Sample
Enrollment: 5479 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
All causes mortality | At discharge, an average of 10 days

SECONDARY OUTCOMES:
All causes mortality | 30 days
adverse cardiovascular and cerebrovascular events (MACCE, death, congestive heart failure, reinfarction and ischemic stroke) | At discharge, an average of 10 days
All causes mortality | 6 months
All causes mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chuanyu Gao, MD, Principal Investigator — Henan Institute of Cardiovascular Epidemiology; Dayi Hu, MD, Principal Investigator — Henan Institute of Cardiovascular Epidemiology
Locations (1):
- Zhengzhou university People's Hospital, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Wang S, Zhang Y, Yang W, Wang X, Zhu Z, Qi D, Zhang J, Zhang J, Gao C. Impact of stress hyperglycemia ratio on incidence of in-hospital cardiogenic shock in patients with ST-elevation myocardial infarction: a prospective, multicenter study. Front Endocrinol (Lausanne). 2025 Dec 12;16:1677084. doi: 10.3389/fendo.2025.1677084. eCollection 2025. PMID 41458546
- [Derived] Wang S, Zhang Y, Qi D, Wang X, Zhu Z, Yang W, Li M, Hu D, Gao C. Development and validation of a risk score for predicting 30-day mortality in patients with ST elevation myocardial infarction. Sci Rep. 2025 Mar 15;15(1):8930. doi: 10.1038/s41598-025-92615-3. PMID 40087520
- [Derived] Zhang Y, Wang S, Cheng Q, Zhang J, Qi D, Wang X, Zhu Z, Li M, Hu D, Gao C; Henan STEMI registry Study Group. Reperfusion strategy and in-hospital outcomes for ST elevation myocardial infarction in secondary and tertiary hospitals in predominantly rural central China: a multicentre, prospective and observational study. BMJ Open. 2021 Dec 20;11(12):e053510. doi: 10.1136/bmjopen-2021-053510. PMID 34930741
- [Derived] Zhang Y, Wang S, Yang S, Yin S, Cheng Q, Li M, Qi D, Wang X, Zhu Z, Zhao L, Hu D, Gao C. Rationale and design of the Henan ST elevation myocardial infarction (STEMI) registry: a regional STEMI project in predominantly rural central China. BMC Cardiovasc Disord. 2019 Nov 28;19(1):271. doi: 10.1186/s12872-019-1250-9. PMID 31783791